CLINICAL TRIAL: NCT05712408
Title: Examining the Impact of an Online, Non-restrictive Diet Among Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-21-629
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet Intervention (Experimental): 8 week non-restrictive diet program
  Interventions: Behavioral: 800g Challenge

INTERVENTIONS:
Behavioral: 800g Challenge — The intervention will involve 8 weeks of an online diet program. Outcomes testing will occur at baseline and post-intervention (following 8 week diet program). During the first 4 weeks, participants will receive educaitonal material and log their daily points in an online application and attend a weekly check-in call with members of the research team. During weeks 5-8, participants will log their daily points in the online application.

SUMMARY:
The current study aims to test an online, non-restrictive diet among persons with multiple sclerosis (MS). Diet is the number one searched second-line therapy among persons with MS, however there are currently no established dietary approaches to improve health and wellbeing among persons with MS. Participants will complete the 8-week diet program using an online application. The primary research question is whether the diet program is acceptable and can improve general health indicators including cholesterol, glucose, body weight, body fat as well as MS symptoms (i.e., walking, cognition, fatigue, and quality of life).

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* a self-reported diagnosis of multiple sclerosis
* relapse free in past 30 days
* non-pregnant
* willing and able to visit University of North Texas on two testing occasions

Exclusion Criteria:

* electronic medical implant, such as a heart pacemaker or an implantable cardioverter defibrillator (ICD)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Metabolic Health | From recruitment to end of 8 week intervention
  Fasted Cholesterol and Gloucose
Body Weight | From recruitment to end of 8 week intervention
  Change in Body Weight
Body Fat | From recruitment to end of 8 week intervention
  Change in Body Fat Percentage

SECONDARY OUTCOMES:
6-Minute Walk | From recruitment to end of 8 week intervention
  Change in 6-Minute Walk Distance
25-Foot Walk | From recruitment to end of 8 week intervention
  Change in 25-Foot Walk Speed
Cognitive Assessments | From recruitment to end of 8 week intervention
  Change in the Brief International Cognitive Assessment in MS Scores. Scores range from 0-208 with higher scores indicating greater cognitive functioning.
Fatigue | From recruitment to end of 8 week intervention
  Change in Fatigue Severity Scale Scores. Scores range from 1-7 with higher scores indicating greater fatigue.
Health-Related Quality of Life | From recruitment to end of 8 week intervention
  Change in SF-12 Scores. Scores range from 0-100 with higher scores indicating greater health-related quality of life.

OTHER OUTCOMES:
Acceptability of Intervention | From recruitment to end of 8 week intervention
  Participants ratings of satisfaction with the diet program. Scores range from 1-5 with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Silveira, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No